CLINICAL TRIAL: NCT00083681
Title: UARK 98-018, A Randomized Phase II Trial of DCEP or DCEP in Combination With Thalidomide as Salvage Therapy for Post Transplantation Relapse in Patients With Multiple Myeloma
Brief Title: DCEP in Combination With Thalidomide as Salvage Therapy for Post Transplantation Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UARK 98-018
Record Dates: First submitted 2004-05-27; First posted 2004-05-28 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Thalidomide; G-CSF; Cisplatin; Etoposide; Dexamethasone; Cytoxan; DCEP; Relapse
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Thalidomide; Dexamethasone; Cyclophosphamide; Etoposide; Cisplatin; Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: Thalidomide
Drug: Dexamethasone
Drug: Cytoxan
Drug: Etoposide
Drug: Cisplatin
Drug: G-CSF

SUMMARY:
The purpose of this investigational trial is to find out how well patients respond and how long their response lasts when treated with a four day chemotherapy regimen involving dexamethasone, cytoxan, etoposide, and cisplatinum, or DCEP with or without thalidomide. Another purpose is to find out what kind of side effects patients will experience.

DETAILED DESCRIPTION:
Each patient enrolled to this study will be assigned to either receive DCEP alone, or in combination with thalidomide. Since it is not known at this time which treatment is the best, you will be placed by chance in one of the two groups.

Treatment consists of three cycles of combination chemotherapy, each over four days. Three drugs, Cytoxan, etoposide, and cisplatin will be given into the vein as a continuous four-day infusion. Decadron will be given by mouth over four days. G-CSF will also be given daily as a shot under the skin to help bone marrow recover.

After 3 cycles of combination chemotherapy, your myeloma will be reassessed. If myeloma is stable or responding, patients will receive an additional 3 cycles of chemotherapy. Then myeloma will again be reassessed and if again found to be stable or responding,3 final cycles of chemotherapy will be given.

Following the completion of chemotherapy, or sooner if your physician feels that the chemotherapy side effects are to great, patients will receive maintenance therapy with dexamethasone. Patients originally assigned to receive thalidomide, will continue to take thalidomide daily throughout protocol treatment.

The major reason for conducting this research is to gather biologic information from patients who have myeloma. Information gained from such research may contribute to a greater understanding of the reasons for treatment failure and may assist in the selection of appropriate treatment for individual patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a confirmed diagnosis of previously treated, active multiple myeloma, with relapse or progression following at least one autologous transplant. High risk is defined as any one of the following at the time of relapse:a) Plasma cell labeling index (PCLI) > 1%, b) Bone marrow plasmacytosis > or = 30%, c)Bartl grade >or = 2 on bone marrow biopsy, or d)Cytogenetic abnormalities of chromosome 13, 11q, or any translocation at the time of relapse.
* Patients must be 18 years of age or older. Women of childbearing age and fertile men must use a medically acceptable means of birth control while on study and for 6 months thereafter.
* Patients must sign an informed consent to participate in this study, and be fully aware of the known teratogenic potential of this drug combination.
* Patients must have a SWOG performance status of 0-2. Patients with a poor performance status (3-4) based solely on bone pain, will be eligible.
* Patients must have adequate renal function, as defined by serum creatinine < or = 3.0 mg/dl
* Before starting treatment, women of childbearing potential should have a negative pregnancy test performed within 24 hours prior to beginning therapy. Written report of a negative pregnancy test must be obtained before a prescription for thalidomide is issued. Pregnancy testing is not required for 1) women wh have been post-menopausal for at least 2 years with no menses, 2) women who have had a hysterectomy.
* Patients must have adequate bone marrow function, as defined by platelet count of 150,000/microliter, unless explained by extensive marrow plasmacytosis.
* Patients must be off chemotherapy (excluding steroids) and local radiotherapy for > 3 weeks prior to entering the study

Exclusion Criteria:

* There must be no evidence of active infection requiring IV antibiotics
* No other concurrent therapy for myeloma is permitted while on protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 1998-06; Study Completion 2005-05

PRIMARY OUTCOMES:
To evaluate the effectiveness of the DCEP chemoregimen with G-CSF support as compared to the DCEP regimen with G-CSF support in combination with thalidomide in high risk patients relapsing after autologous transplantation.

SECONDARY OUTCOMES:
To evaluate the quantitative and qualitative toxicities associated with the regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Fassas, M.D., Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences/MIRT, Little Rock, Arkansas, United States

REFERENCES:
- See also: Myeloma Institute for Research & Therapy website — http://myeloma.uams.edu